CLINICAL TRIAL: NCT02137876
Title: Effects of Thymoglobulin on Proliferation, Activation, and Differentiation of Human B Cells
Brief Title: Effects of Thymoglobulin on Human B Cells
Status: Withdrawn | Type: Observational
Why Stopped: Subject recruitment was unsuccessful.
Sponsor: Northwestern University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Lorenzo Gallon, Professor, Northwestern University
Other Study IDs: STU00092183
Record Dates: First submitted 2014-04-30; First posted 2014-05-14 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acute Humoral Rejections; Chronic Humoral Rejections; Transplant
Keywords: B cells; Thymoglubulin; humoral rejections; transplant; rATG
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20ml of whole blood will be drawn from each subject each time they are asked to have blood drawn. The total amount of blood collected from subjects will not exceed 360 ml (1.5 cups) within any eight week period throughout the two year timespan patients may be asked to participate in this study.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood Draws — Patients will be asked to provide blood for immune tests.Patients will not take any study medications, all the research will be performed on blood donated for the study.Patients will donate about 20mls of blood (2 tbls)to be used to determine the subject's blood group and tissue typing (genetic).Results and the patient's contact information will be maintained in a database that is accessible only by the investigators and study personnel conducting the study.For the duration of this study, the investigator will contact patients by phone to request additional samples when needed. Study staff may ask patients donate more blood on short notice (1 day). This will consist of 60-120 ml (6-12 tbls) of blood.The frequency of blood collection will not exceed more than 2 times per week.The total amount of blood collected from subjects will not exceed 360 ml (1.5 cups) within any eight week period throughout the two year timespan patients may be asked to participate in this study.

SUMMARY:
This study is being done to better understand how immunosuppressive medications (anti-rejection medications that may or may not be approved by the Food and Drug Administration (FDA)) affect the alloimmune response (how a person's immune system reacts against another person's immune system). This will be determined by the blood tests run on the patients donated blood cells.

Specifically, the investigators will test different immunosuppression medications using in-vitro assays (in the laboratory, in test tubes) alone and/or in combination to test how they can affect B-cell proliferation and differentiation, leading to an altered distribution among defined B-cell subsets and to study if exposure of B cells to thymoglobulin can have effects on subsequent interaction between B and T cell in vitro.

To enable the investigators to understand how immunosuppressant medications affect immune systems in transplant patients, the investigators need to understand how they affect immune systems in healthy people. To do this, the investigators will need to study blood collected from healthy volunteers.

DETAILED DESCRIPTION:
This is a research study of healthy subjects who will furnish blood samples for various assays over a period of one year.

Peripheral blood mononuclear cells (PBMC) will be isolated from healthy volunteers and CD19+ B cells will be selected using CD19 magnetic micro-beads.

B-cell cultures will be performed in culture medium consisting of Iscove's MDM (IMDM) medium (Gibco, Paisley, UK) supplemented with 10% human serum (HNS- GemCell), 0.5 ml Human Insulin (Sigma), 200mM L-Glutamine (Sigma) and 0.5% Gentamycin (Gibco).

Total CD19+B cells will be cultured in the presence of anti-IgM (3μg/ml), anti-CD40 (100ng/ml), IL-21 (100ng/ml) (BCR/CD40-stimulation) for 6 days in culture plates 96 wells round bottom (1.0x105 cells/well), and Thymoglobulin at different concentrations (10 to 100 μg/ml) with or without calcineurin inhibitor (Tacrolimus, TAC) and mTOR inhibitor (Sirolimus, SRL) will be added at day 0.

A variety of parameters of B cell activity including proliferation, activation, differentiation and cytokine production will be monitored by flow cytometry.These experiments are further explained in the outcome measures section below.

The investigators will conduct univariate and bivariate analyses for all variables. The investigators will evaluate continuous variables using t-tests or F-tests and categorical variables using Chi-square or Fisher Exact tests. The investigators will examine data distributions and test all variables for linear relationships or non-linear relationships. Descriptive statistics (means, standard deviation, frequency) and correlations (both Pearson and Spearman) among variables will be conducted to assess the data. Necessary transformation and imputations will be conducted based on the raw data distribution. All data analyses will be performed using SAS 9.3 statistical software (SAS Inc., Cary, NC). All tests will be two-sided and an error rate of α <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

The patient:

1. should be more than 18 years old,
2. should weigh more than 110 lbs and
3. should not be pregnant at the time of blood donation.

Exclusion Criteria:

(1) Not fitting within inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will consist of healthy volunteers who meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
CD19+B cell division | 12 days
  3-6x106 cells of interest will be labeled with 1.5μM CFSE before stimulation. After 6 days, B cells will be recovered, washed, counted and used to define marker settings. The cell phenotype will be analyzed by five-color flow cytometry (FC500, Beckman-Coulter) and by 13-color flow cytometry (Fortessa) and data will be analyzed using CXP software. The supernatant of these B-cell cultures will be using for the cytokines detection, and to determine the number of IgM and IgG producing cells by Luminex.At day 6, cells will be re-stimulated with phorbol 12-myristate 13-acetate (PMA) and Ionomycin, and analyzed by intracellular cytokine staining. Total CD19+ B cells will be sorted into a CD27- (naïve) and CD27+ (memory) B-cell fraction and the phenotypic characterization (assessed by flow cytometry) of these cells will be showed after 6 days of culture with anti-IgM (5μg/ml), anti-CD40 (100ng/ml), and IL-21 (100ng/ml) in the presence or absence of the drugs.

SECONDARY OUTCOMES:
proliferated T-cells | 6 days
  The investigators will co-culture B cells (pre-stimulated with α-IgM and α-CD40 mAb plus IL-21 for 6 days in the presence and absence of Thymoglobulin) with allo-CD4+CD25- T cells (ratio 2:1). After 6 days the investigators will analyze the % of proliferated T-cells and the cytokine production.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Comprehensive Transplant Center, Chicago, Illinois, United States